CLINICAL TRIAL: NCT03607292
Title: A Comparison Of Block Quality In Anterior And Posterior Approach To Sciatic Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Abdulkadir Yektas, Principal Investigator, Bagcilar Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sciatic Nerve Block
Record Dates: First submitted 2018-06-11; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Ankle Fractures
Keywords: Sciatic Nerve Blocks; Ankle surgery
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Intervention Model Description: Randomize, single blind, prospective
Masking Description: A single blinded anesthesiologist performed posterior or anterior sciatic nerve block and femoral block and left the operating room 'after the nerve block was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Anterior sciatic nerve block
  Interventions: Procedure: Anterior sciatic nerve block
- Group P (Experimental): Posterior sciatic nerve block
  Interventions: Procedure: Posterior sciatic nerve block

INTERVENTIONS:
Procedure: Anterior sciatic nerve block — A straight line along the femoral catheter was drawn between the anterior superior iliac spine and the finger palpating the pubic bone, the index finger was placed over the femoral artery pulse, a line was drawn perpendicular to the femoral fold. Over the pulse of the femoral artery, a point 4-5 cm lateral. The sciatic nerve was imaged by USG along the needle route and the needle was advanced to the nerve.
  Arms: Group A
Procedure: Posterior sciatic nerve block — Patient was positioned laterally, with the limb to be blocked uppermost. The lower leg was straight extended and the upper extremity was bent 90° from the knee and was directed forward on the lower straight extended extremity. The patient's greater trochanter and posterior superior iliac spine were palpated and joined with a line, and a line was drawn 4 cm above the first line perpendicular to the caudal line. The USG probe was placed between the greater trochanter and the coccyx at the entry point of the needle and the needle was advanced by imaging the nerve.
  Arms: Group P

SUMMARY:
Co-administration of the sciatic nerve block and femoral nerve block may provide anesthesia and analgesia in patients undergoing lower extremity surgery. Several approaches to sciatic nerve block have been described. The anterior and posterior approaches are two of the approaches used to make the sciatic nerve block. In our study, n = 20 patients for Group A and n = 25 patients for Group P were included. Then, sciatic nerve block and femoral nerve block were performed to each patient by using anterior or posterior approach randomly. After the block is performed, the sensory and motor block start and end times, the first intraoperative fentanyl requirement time and total amount of fentanyl required, the first Diclofenac sodium requirement time, and the total amount of diclofenac sodium that patients required were determined. As the groups were compared to each other; the time to start sensory block was statistically significantly lower, the first fentanyl requirement time was statistically significantly earlier and the total amount of fentanyl required was statistically significantly lower in Group P. Patient satisfaction, anesthesia quality and surgical quality were statistically significantly higher in Group P. In this study, the investigators concluded that if a patient does not have pain secondary to fracture, posterior approach to sciatic nerve block can be performed, whereas, if a patient has pain secondary to fracture, anterior approach to sciatic nerve block can be performed in order to avoid repositioning.

DETAILED DESCRIPTION:
Forty five patients were enrolled to the study. These patients were classified in the American Society of Anesthesiologists (ASA) I-II group. The written informed consent of each patient was obtained.

The study was randomized, single blinded and prospectively planned. Randomization was done according to the randomization table prepared by the computer. A single blinded anesthesiologist performed posterior or anterior sciatic nerve block and femoral block and left the operating room after the patient was corrected after the nerve block was completed and another anesthesiologist followed the patient without knowing what approach was used. Before initiating the study, the required number of participants was determined according to the results of a pilot study which was performed by enrolling 10 patients in each group.

The time of sciatic nerve sensory block onset ± Standard Deviation (SD) was calculated as 8,88 ± 4,87 minutes for Group A (anterior approach to sciatic nerve block + femoral nerve block) and 4.70 ± 2.05 minutes for Group P (posterior approach to sciatic nerve block + femoral nerve block). The sample size was calculated on websites named www.power and www.sample size.com/Calculators/Compare-2-means/2-Sample-Equality. The sample size was calculated as 25 (n = 25) for Group A and 7 (n = 7) for Group P, while α = 5% with 85% power. Whereas, 20 patients were enrolled for Group P because small n should be greater than half of large n for reliability.

The patient's age, gender, height, weight, other existing diseases, drug use, smoking history, anesthetic method applied, operation time, tourniquet time, ASA classification, intraoperative first fentanyl requirement time and total fentanyl amount during the operation, measurements of systolic, diastolic and mean blood pressures, heart rate and peripheral oxygen saturation values before and after the block, motor and sensory block start and end times after sciatic and femoral block were performed, first Diclofenac sodium time and total Diclofenac sodium amount administered in 24 hours, visual analogue scale (VAS) values, patient satisfaction, anesthetic quality from the point of anesthesiologist, and surgical quality from the point of surgeon were recorded.

Patients who were informed about VAS one day before and not administered premedication were taken to the regional block room and routine electrocardiogram, noninvasive arterial blood pressure and peripheral pulse oximeter monitoring were performed. Baseline values of blood pressure, heart rate and peripheral oxygen saturation were recorded before the block was performed. During the operation these values were recorded every 5 minutes.

First of all, the sciatic nerve block with anterior approach was performed in the group A. The block was performed by the needle named Stimuplex® A (21G 0.80-150), which was at 30 ° and isolated in conjunction with a block nerve stimulator (Stimuplex HNS nerve stimulator BRAUN, Germany) and ultrasonography (USG) (Diagnostic ultrasound system, Model SDU 450 XL Class-1 type B Shimadzu Corporation, Japan) mm). A total of 40 ml of a local anesthetic solution composed of 30 ml of 0.5% isobaric bupivacaine and 10 mL of 2% lidocaine was prepared.

In both the anterior and posterior approach to sciatic nerve block and the femoral nerve block, nerve stimulation was done with a frequency of 2 Hz and with 1 Milliampere (mA) current, and the stimulus intensity was gradually reduced to 0.4 mA as long as the as response was obtained. Femoral nerve block: The nerve was visualized in direct USG coincidence and the needle was oriented to the nerve. After the contraction of vastus medialis, vastus intermedius, and vastus lateralis muscles were visualized, local anesthetic mixture of 20 ml was injected and dissemination of the local anesthetic solution was imaged by USG (Linear probe).

Anterior sciatic nerve block: Technically, a straight line along the femoral catheter was drawn between the anterior superior iliac spine and the finger palpating the pubic bone, the index finger was placed over the femoral artery pulse, a line was drawn perpendicular to the femoral fold. Over the pulse of the femoral artery, a point 4-5 cm lateral to this line was marked and this point was identified as the needle entry point. The sciatic nerve was imaged by USG (Convex probe) along the needle route and the needle was advanced to the nerve. When the plantar flexion, dorsal flexion and eversion of the foot were observed, 20 mL of local anesthetic mixture was given and local anesthetic spread was imaged by USG simultaneously.

Posterior sciatic nerve block: The patient was positioned laterally, with the limb to be blocked uppermost. The lower leg was straight extended and the upper extremity was bent 90 ° from the knee and was directed forward on the lower straight extended extremity. The patient's greater trochanter and posterior superior iliac spine were palpated and joined with a line, then the middle point of this line was found and a line was drawn 4 cm above the first line perpendicular to the caudal line. The end point of the 2nd line was taken as the entry point of the needle. The USG probe was placed between the greater trochanter and the coccyx at the entry point of the needle and the needle was advanced by imaging the nerve. When the plantar flexion, dorsal flexion, and eversion of the foot were observed, 20 mL of local anesthetic mixture was given and local anesthetic spread was imaged by USG simultaneously.

After the blocks were completed, the motor block was assessed by monitoring the movement of the ankle joint and knee, and sensory block was assessed with a cold application every minute, and the block start times were recorded. When the patient was not receiving any stimulation with cold application on sciatic and femoral stimulation areas, it was recorded as the start time of the full femoral-sciatic sensory block. When the knee joint could not be moved at all, it was recorded as the start time of the full femoral motor block.

When the ankle joint was unable to move, it was recorded as the start time of the full sciatic motor block. After the block was fully achieved, the tourniquet was applied to the extremity to be operated and was inflated. Patients underwent surgery 30 minutes after the block was provided. After the surgical procedure started, 1 μg kg-1 fentanyl was injected intramuscularly when the VAS values of the patients were greater than 4. The patient's first fentanyl requirement time and the total amount of fentanyl administered during the operation were recorded.

When the arterial blood pressures of a patient fell below 80% of pre-block values, 5 mg ephedrine was administered intramuscularly. Intravenous administration of 0.5 mg atropine was planned when the heart rate dropped below 50 beats min-1. When the patients had nausea and vomiting, 4 mg of ondansetron (Zofer, Adeka, Turkey) was administered intramuscularly.

After the operation was completed, the patients were taken to the postoperative care unit. Patients were followed in the postoperative care unit until the block was completely terminated. Patients were sent to the clinic after the block was terminated. The time of first diclofenac sodium required by the patients and the amount of diclofenac sodium administered within 24 hours of the post-operative period were recorded. The first postoperative diclofenac sodium dose was administered when a patient had VAS values of 4 or more.

All data were evaluated using the SPSS 11.5 for Windows package program. The normality distribution of the data was assessed by the Kolmogorov-Smirnov test. In the complementary statistics of the data, the mean ± standard deviation values for the parametric tests and the median (minimum-maximum) for the nonparametric tests were used. Categorical data were given as %n. Independent-Samples T Test was used for binary comparison of the data of the groups, chi-square test was used for comparing the categorical data of the groups. In order to make comparison in all of the statistical data, p <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were between the ages of 18 to 65 and were going to be operated due to lateral and/or medial malleolus fracture.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2014-03-18 (Actual); Study Completion 2014-12-20 (Actual)

PRIMARY OUTCOMES:
Comparison of sensorial block start time after sciatic nerve block performed with anterior and posterior approaches. | up to 20 minutes.
  Sensory block was assessed with a cold application every minute, and the block start time was recorded. When the patient was not receiving any stimulation with cold application on sciatic stimulation area, it was recorded as the start time of the full sciatic sensory block.

SECONDARY OUTCOMES:
Comparison of sensorial block end time after sciatic nerve block performed with anterior and posterior approaches. | up to 300 minutes.
  Sensory block was assessed with a cold application every minute, and the block end time was recorded. When the patient received any stimulation with cold application on sciatic stimulation area, it was recorded as the end time of the full sciatic sensory block.
Comparison of sensorial block start time after femoral nerve block performed with anterior and posterior approaches. | up to 20 minutes.
  Sensory block was assessed with a cold application every minute, and the block start time was recorded. When the patient was not receiving any stimulation with cold application on femoral stimulation area, it was recorded as the start time of the full femoral sensory block.
Comparison of sensorial block end time after femoral nerve block performed with anterior and posterior approaches. | up to 160 minutes.
  Sensory block was assessed with a cold application every minute, and the block end time was recorded. When the patient received any stimulation with cold application on femoral stimulation area, it was recorded as the end time of the full femoral sensory block.
Comparison of patient satisfaction | After surgery up to 24 hours.
  Patient satisfaction:0: failed,1: weak, 2: moderate, 3: good, 4: excellent
Comparison of anesthesia quality in groups | After surgery up to 24 hours.
  Anesthesia quality assesment by Anesthesiologist; 1: Failed; general anesthesia was required, 2: Moderate, complainant, complementary analgesic was needed, 3: Good, little complainant, no need for complementary analgesia, 4: Excellent, patients do not complain
Comparison of surgical quality in groups | After surgery up to 24 hours.
  surgical quality assesment by Surgeon; 1: Failed; general anesthesia was required, 2: Moderate, complainant, complementary analgesic was needed, 3: Good, little complainant, no need for complementary analgesia, 4: Excellent, patients do not complain
Comparison of intra-operatively administered total fentanyl amount and total diclofenac sodium amount in the postoperative first 24-hour periods in the group. | within 24 hours of the post-operative period
  After the surgical procedure started, 1 μg kg-1 fentanyl was injected intramuscularly when the VAS values of the patients were greater than 4. The patient's total amount of fentanyl administered during the operation was recorded. After the operation was completed, the amount of diclofenac sodium administered within 24 hours of the post-operative period were recorded.
Comparison of intra-operatively administered first fentanyl requirement time and first diclofenac sodium requirement times in the postoperative first 24-hour periods in the groups. | within 24 hours of the post-operative period
  After the surgical procedure started, 1 μg kg-1 fentanyl was injected intramuscularly when the VAS values of the patients were greater than 4. The patient's first fentanyl requirement time during the operation were recorded. After the operation was completed, the time of first diclofenac sodium required by the patients within 24 hours of the post-operative period was recorded. The first postoperative diclofenac sodium dose was administered when a patient had VAS values of 4 or more.
Comparison of motor block start time after sciatic nerve block performed with anterior and posterior approaches. | every minute up to 20 minutes.
  When the ankle joint was unable to move, it was recorded as the start time of the full sciatic motor block.
Comparison of motor block end time after sciatic nerve block performed with anterior and posterior approaches. | every minute up to 160 minutes.
  When the ankle joint was able to move, it was recorded as the end time of the full sciatic motor block.
Comparison of motor block start time after femoral nerve block performed with anterior and posterior approaches. | every minute up to 20 minutes.
  When the knee joint could not be moved at all, it was recorded as the start time of the full femoral motor block.
Comparison of motor block end time after femoral nerve block performed with anterior and posterior approaches. | every minute up to 110 minutes.
  When the knee joint could be moved at all, it was recorded as the end time of the full femoral motor block.